CLINICAL TRIAL: NCT03496350
Title: Culturally Adapted Transdiagnostic Internet-delivered Cognitive Behavioural Therapy in Arabic for Anxiety and Depression
Brief Title: Internet-delivered Cognitive Behavioural Therapy in Arabic for Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHA
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants get randomly assigned to either treatment or wait-list control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet CBT (Experimental): Internet-based cognitive behavioural therapy in Arabic with therapeutic guidance through email.
  Interventions: Behavioral: Internet-delivered CBT
- Wait-list (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: Internet-delivered CBT — Culturally adapted transdiagnostic internet-delivered CBT in Arabic
  Arms: Internet CBT

SUMMARY:
The purpose of this study is to evaluate the efficacy of a culturally adapted internet-administrated cognitive behaviour therapy (ICBT) in Arabic for anxiety and depression

DETAILED DESCRIPTION:
The study will compare the effect of the intervention against a wait-list control. The intervention tested is based on cognitive behavior therapy delivered over the internet via a secure treatment platform. Participants in the study are recruited from the general public via social media. The intervention is in Arabic.

ELIGIBILITY:
Inclusion Criteria:

* Be above 18 years of age
* Have symptoms of anxiety and/or depression
* Be able to read and write in Arabic
* Have access to computer or smartphone

Exclusion Criteria:

* Suicidal ideation
* Alcohol addiction
* Other major primary psychiatric disorder
* Ongoing psychological treatment
* Recent (during last 4 weeks) change in psychiatric medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | pre-treatment ,week 3, week 6, week 8 and 12 months post-treatment
  The PHQ-9 is a nine-item self-report questionnaire that measures symptoms of depression. It is scored from 0-27 with a higher score reflecting more severe symptoms.
Change in Generalised Anxiety Disorder-7-item scale, (GAD-7) | pre-treatment ,week 3, week 6, week 8 and 12 months post-treatment
  The GAD-7 is a seven-item self-report questionnaire that measures symptoms of anxiety. It is scored from 0-21 with a higher score reflecting more severe symptoms.

SECONDARY OUTCOMES:
Alcohol Use Disorder Identification Test (AUDIT) | pre-treatment, week 8
  Measures alcohol consumption, drinking behaviors, and alcohol-related problems. It is scored from 0-40 with higher scores reflecting more alcohol consumption, drinking behaviors, and alcohol-related problems.
Insomnia Severity Index (ISI) | pre-treatment, week 8
  Self-reported symptoms of insomnia. It is scored from 0-28 with higher scores reflecting more symptoms of insomnia.
Impact of Events Scale - Revised (IES-R) | pre-treatment, week 8
  Self-reported symptoms of post-traumatic stress. It is scored from 0-88 where higher scores reflect more symptoms.
Perceived Stress Scale (PSS) | pre-treatment, week 8
  Self-reported stress-related symptoms. It is scored from 0-56 with higher scores reflecting more symtoms of perceived stress.
"Brunnsviken Brief Quality of Life Scale" (BBQ) | pre-treatment, week 8
  Self-reported quality of life. The scale is scored from 0-96 with a higher score reflecting higher self-reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No